CLINICAL TRIAL: NCT06861504
Title: The Femscope Calm Collect Device to Obtain Cervical Cells for Cancer Screening
Brief Title: The Femscope Calm Collect Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Marilyn S Filter, Professor of Nursing, School of Nursing, The University of Michigan-Flint, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HUM00224241
Record Dates: First submitted 2025-01-10; First posted 2025-03-06 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-10

CONDITIONS: Cervical Cancer
Keywords: Cervical cancer screening
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Intervention Model Description: The Femscope Calm Collect Device will be used to collect a sample of cervical cells that a board-certified pathologist will read.
Masking Description: All specimens collected will receive a randomized number so the pathologist is not aware of the samples collected by the traditional brush method (Pap smear) and the cells collected by the Femscope Calm Collect Device.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Cervical cell collection of traditional brush and Femscope Calm Collect Device (Experimental): Cervical cells of the Femscope Calm Collect Device will be evaluated by a board-certified pathologist to determine if the quality and quantity of cells are equivalent to the traditional brush collection.
  Interventions: Device: Femscope Calm Collect Device

INTERVENTIONS:
Device: Femscope Calm Collect Device — The Femscope Calm Collect Device uses a patented brush for cervical cell collection.

SUMMARY:
The goal of this clinical trial is to determine if cervical cells collected by the Femscope Calm Collect Device in women (sex assigned at birth) of adult age are the same quality and quantity as the cervical cells collected by the traditional brush method for cervical cancer screening. The main questions it aims to answer are:

1. Increase the number of women who get screened for cervical cancer.
2. Improve patient acceptance of getting cervical screening on a routine basis.
3. Decrease pain and discomfort for patients having a PAP smear procedure.

Participants will

* Have two vaginal exams to collect cervical cells.
* State decreased pain and discomfort for patients having a PAP smear procedure.
* The Femscope Calm Collect Device (FCCD) will be more comfortable for the patient as measured by a patient satisfaction survey comparing the FCCD and the traditional speculum method of obtaining cervical cells.

DETAILED DESCRIPTION:
The FemScope Calm Collect Device is a novel medical device intended for vaginal inspection, cervical cancer screening, rectal cancer screening, and discharge/cell retrieval. The device allows for increased comfort (emotionally and physically) to the patient while meeting the requirements of a genital exam.

The FemScope system includes a light and camera, enabling visualization of the vagina and cervix and display on a screen. It also provides brushing/retrieval means, allowing the provider to obtain necessary cervical cells for a pap smear, HPV, and specimens needed for sexually transmitted disease (STI) testing. The system will also allow the direct visualization of rectal tissue sampled for human papillomavirus/rectal cancer. The system is designed to replace the speculum, provide the tools needed to perform comprehensive pelvic and topical rectal exams, provide cervical cancer screens, and be cost-competitive with existing speculum and tissue swab systems. It is simple and easy to use. The device comprises a reusable base portion, a removable protective sleeve, and a single-use cell retrieval cap for improved cost-effectiveness.

This instrument will revolutionize women's health care, replacing the antiquated speculum examination with modern scopes like those used to visualize many other portions of the human body. Having the instrument designed to facilitate exams in the LGBTQIA community is sorely needed and will improve gynecologic and genital examinations in that community

ELIGIBILITY:
Inclusion Criteria:

- Healthy female ages 21-45 with female reproductive organs present at the time of study.

Exclusion Criteria:

* Pregnancy
* Menopausal
* Age less than 21 years
* Age of 46+ years
* History of reproductive cancer
* Hysterectomy

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — All participants must have female sexual organs present at birth.
Enrollment: 13 (Actual)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Specimen Adequacy Using The Femscope Calm Collect Device vs. The Traditional Brush Method | 1 hour
  Specimen adequacy will be assessed using the Bethesda System For Reporting Cervical Cytology. Specimens will be rated as Satisfactory or Unsatisfactory for evaluation. The presence/absence of a Endocervical/Transformation Zone (EC/TZ) component, partially obscuring blood, and inflammation are indicators the Pap test is satisfactory for evaluation.
Number of Participants Who Experienced Pain/Discomfort During The Femscope Calm Collect Procedure | Immediately post-procedure
  A binary (yes/no) assessment of whether the participant experienced pain or discomfort during the Femscope Calm Collect Procedure.
Number of Participants Who Experienced Pain/Discomfort During The Regular Pap Procedure | Immediately post-procedure
  A binary (yes/no) assessment of whether the participant experienced pain or discomfort during the regular Pap procedure

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan Flint, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Will need to determine if Femscope Calm Collect Device meets cervical cell collection criteria.
Supporting Information: Study Protocol, CSR
Time Frame: 1/1/2026
Access Criteria: Research team